CLINICAL TRIAL: NCT05850507
Title: A Randomized, Double-blind, Active-controlled Clinical Study Evaluating the Immunogenicity and Safety of Omicron BA.4/5-Delta Strain Recombinant Novel Coronavirus Protein Vaccine (CHO Cells) in People 18 Years of Age and Older
Brief Title: Omicron BA.4/5-Delta Strain Recombinant Novel Coronavirus Protein Vaccine (CHO Cells)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LKM-2023-NCV-02
Record Dates: First submitted 2023-04-07; First posted 2023-05-09 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2023-05

CONDITIONS: Coronavirus
Keywords: Omicron BA.4/5-Delta strain
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Intramuscular injection of 25μg/0.5ml Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cells) in the deltoid muscle of the upper arm.
  Interventions: Biological: Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cells)
- Control group (Active Comparator): Intramuscular injection of 25 μg/0.5 ml recombinant novel coronavirus protein vaccine (CHO cells) into the deltoid muscle of the upper arm.
  Interventions: Biological: Recombinant novel coronavirus protein vaccine (CHO cells)

INTERVENTIONS:
Biological: Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cells) — Intramuscular injection of deltoid muscle of upper arm of 25μg/0.5ml/person dose Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cells).
  Arms: Study Group
Biological: Recombinant novel coronavirus protein vaccine (CHO cells) — Intramuscular injection of deltoid muscle of upper arm of 25μg/0.5ml/person dose Recombinant new coronavirus vaccine (CHO cells) .
  Arms: Control group

SUMMARY:
Popular title: Clinical study of Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cells).

Purpose of the study: Main objectives: To evaluate the immunogenicity and safety of Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cells) against the new coronavirus prototype strain and Omicron variant (BA.5, BF.7) after vaccination in people aged 18 years and older. Secondary purposes: To evaluate the immune persistence of Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cells) against the new coronavirus prototype strain and Omicron variant (BA.5, BF.7) after vaccination in people aged 18 years and older.

Overall design: Studies were randomized, double-blind, active, controlled study design.

Study group: people aged 18 years and above who have completed primary immunization or booster immunization of the new coronavirus vaccine for more than 6 months.

Study group: Randomly divided into study group and control group according to the 1:1 ratio, of which 225 subjects in the study group and 225 subjects in the control group were vaccinated with study vaccine and control vaccine respectively.

DETAILED DESCRIPTION:
Popular title: Clinical study of Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cells). Research vaccine: Name: Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cell), main components: receptor binding region (OD-RBD) protein (25μg/0.5mL) of novel coronavirus spike glycoprotein, aluminum hydroxide adjuvant. Control vaccine: Name: Recombinant novel coronavirus protein vaccine (CHO cells), main components: receptor-binding region (NCP-RBD) protein (25μg/0.5mL) of novel coronavirus spike glycoprotein, aluminum hydroxide adjuvant. Indications: Prevention of respiratory diseases caused by novel coronavirus infection Research population: healthy people ≥60 years old Research institution: Yijishan Hospital, Wannan Medical College Research Objective: Main objective: To evaluate the immunogenicity and safety of Omicron BA.4/5-Delta recombinant novel coronavirus protein vaccine (CHO cells) against the prototype strain of the new coronavirus and Omicron variant (BA.5, BF.7) after vaccination in people aged 18 years and above.

Secondary objective: To evaluate the immune persistence of Omicron BA.4/5-Delta strain recombinant novel coronavirus protein vaccine (CHO cells) against the new coronavirus prototype strain and Omicron variant (BA.5, BF.7) after vaccination in people aged 18 years and above.

Research Plan: Sample size: Based on the efficacy test of the experimental group against the new coronavirus Omicron strain BA.4/5 and the control group against the new coronavirus Omicron strain BA.4/5 free neutralizing antibody GMC, the standard deviation of the antibody level after logarithmic conversion with base 10 is assumed to be σ = 0.65. With an overall power of 90%, a class I error of 0.025 on one side, a 95% confidence interval lower bound of the GMC ratio >1, and an expected GMC ratio of 2.1, 81 cases are required for each group. In summary, considering about 15% shedding, the sample size of the experimental group and the control group was allocated 1:1, that is, 100 cases were needed in each group, and a total of 200 cases were needed. At the same time, according to the guiding principles, in order to observe the safety of the test seedlings, the total sample size was expanded to 450 cases, that is, 225 cases were required for the experimental group and the control group.

Study group: The study plans to recruit 450 cases of people aged 18 and above who have completed the basic immunization or booster immunization of the new coronavirus vaccine for more than 6 months, and are randomly divided into the research group and the control group according to the ratio of 1:1, of which 225 subjects in the research group and 225 subjects in the control group are vaccinated with the study vaccine and the control vaccine respectively. The 450 participants should include 150 elderly (60 years and older) and 300 adults (18-59 years old).This clinical trial will set up immunogenic subgroups in the enrolled 450 patients, a total of 200 cases, including 100 cases in the study group and 100 cases in the control group. All subjects were tested for neutralizing antibody immunogenicity (BA.5 strain) in pre-neutralizing serum, and the first 100 subjects in the study group and control group were included in the immunogenicity subgroup in order of study number. If there are less than 100 neutralizing antibody negative subjects in the study group or control group, the immunogenic subgroup of neutralizing antibody positive subjects will be included in the immunogenic subgroup of neutralizing antibody positive subjects in the order of study number until the number reaches 100.

Safety endpoints:

1. Incidence of all AEs within 30 days of vaccination:

1. incidence of total AE ;
2. the incidence of AEs associated with the study vaccine ;
3. Grade 3 and above AE incidence ;
4. incidence of grade 3 and above AEs associated with the investigational vaccine ;
5. the incidence of AE leading to withdrawal ;
6. The incidence of AEs leading to withdrawal associated with the study vaccine. Incidence of all serious adverse events (SAEs), vaccine-related SAEs within 6 months after vaccination.

Immunogenicity endpoint: Primary endpoint:

Geometric mean titer (GMT) and positive conversion rate of neutralizing antibodies against the Omicron variant (BA.5) of the novel coronavirus in the study and control groups 14 days after the immunogenicity subgroup received the investigational vaccine.

Secondary endpoints:

1. 14 days after the immunogenic subgroup of subjects received the investigational vaccine, the neutralizing antibody GMT, growth multiple (GMI), and positive conversion rate of the research group and the control group against the new coronavirus prototype strain and the Omicron variant (BF.7);
2. 14 days after the immunogenicity subgroup of subjects received the investigational vaccine, the neutralizing antibody GMI of the research group and the control group against the new coronavirus Omicron variant (BA.5);
3. 6 months after the immunogenicity subgroup received the investigational vaccine, the neutralizing antibody GMT, GMI, and positive conversion rate of the study group and the control group against the new coronavirus prototype strain and Omicron variant (BA.5, BF.7).

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years of age or older at the time of signing the informed consent form;
2. The subject himself voluntarily participates in the study, signs the informed consent form, and can provide legal identification, understand and comply with the requirements of the research protocol;
3. More than 6 months after completing the basic immunization or booster immunization of the new coronavirus vaccine; Female subjects of childbearing age and male subjects who were able to use effective contraception during the study.

Exclusion Criteria:

Participants were not eligible for study if they had any of the following:

1. Previous history of severe allergy to any vaccine, or history of severe allergy to any component of the study vaccine, including aluminum preparations, such as: anaphylactic shock, allergic laryngeal edema, Henoch-Schönlein purpura, thrombocytopenic purpura, dyspnea, angioedema, allergic constitution (such as allergy to two or more drugs, food or pollen), etc.;
2. fever (axillary body temperature≥ 37.3°C) within 72 hours before enrollment, or axillary body temperature ≥ 37.3°C on the day of enrollment;
3. Patients infected with the new coronavirus within 3 months before enrollment (asymptomatic infection or positive nucleic acid or antigen test of the new coronavirus);
4. Patients with aplastic anemia that has not been relieved, primary immune thrombocytopenia (ITP) active period, and uncontrolled coagulation diseases;
5. history of congenital or acquired immunodeficiency or autoimmune disease; no history of spleen or spleen surgery or trauma; or receive immunomodulators within 6 months, such as corticosteroids in immunosuppressant doses (dose reference: equivalent to prednisone 20 mg/day for more than one week); or monoclonal antibodies; or thymus peptide; or interferon, etc.; However, topical medications (such as ointments, eye drops, inhalers, or nasal sprays) are allowed; Lymphoproliferative disorders are not controlled;
6. Non-live vaccine ≤ 14 days before vaccination and live attenuated vaccine 30 days before ≤vaccination;
7. Patients with malignant tumors who are undergoing chemotherapy, radiotherapy, immunotherapy, etc. before and after surgery; Patients in the state of organ transplantation;
8. Those suffering from uncontrolled epilepsy and other progressive neurological diseases (such as transverse myelitis, Guillain-Barre syndrome, demyelinating diseases, etc.);
9. Patients with acute diseases, or acute exacerbations of chronic diseases, or uncontrolled severe chronic diseases, such as hypertension that cannot be controlled by drugs (systolic blood pressure ≥ 160mmHg and/or diastolic blood pressure ≥100mmHg);
10. Lactating women or pregnant women; The investigator believes that the participant has any disease or condition that would put the participant at risk, the participant cannot complete the study as required by the protocol, and there are circumstances that interfere with the assessment of vaccine response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
The number of adverse events after intramuscular injection | 6 months after vaccination
  The observation of adverse events mainly come from vital sign detection and laboratory examination (including blood routine/urine routine/blood biochemistry/electrocardiogram and chest X-ray), local reactions and systemic reactions after injection.
Laboratory markers of immunity | 14 days after vaccination
  Geometric mean titer (GMT) of neutralizing antibodies against the Omicron variant (BA.5) after vaccination with the investigational vaccine.
Immunogenic end points | 14 days after vaccination
  Positive conversion rate of the Omicron variant (BA.5) of the new coronavirus after vaccination with the investigational vaccine.

SECONDARY OUTCOMES:
Laboratory markers of immunity | 14 days after vaccination
  Geometric mean titer (GMT) of neutralizing antibodies against the prototype strain of the new coronavirus, Omicron variant (BF.7) after vaccination with the investigational vaccine.
Laboratory markers of immunity | 14 days after vaccination
  Growth multiple (GMI) of the new coronavirus prototype strain and Omicron variant (BF.7) after vaccination with the investigational vaccine.
Immunogenic end points | 14 days after vaccination
  Positive conversion rate against the prototype strain of the new coronavirus, Omicron variant (BF.7) after vaccination with the investigational vaccine.
Laboratory markers of immunity | 14 days after vaccination
  Growth multiple (GMI) of the new coronavirus prototype strain and Omicron variant (BA.5) after vaccination with the investigational vaccine.
Laboratory markers of immunity | 6 months after vaccination
  Geometric mean titer (GMT) of neutralizing antibodies against the prototype strain of the new coronavirus, Omicron variant (BA.5, BF.7) after vaccination with the investigational vaccine.
Laboratory markers of immunity | 6 months after vaccination
  Growth multiple (GMI) of the new coronavirus prototype strain and Omicron variant (BA.5, BF.7) after vaccination with the investigational vaccine.
Immunogenic end points | 6 months after vaccination
  Positive conversion rate against the prototype strain of the new coronavirus and the Omicron variant (BA.5, BF.7) after vaccination with the investigational vaccine.

CONTACTS AND LOCATIONS:
Locations (1):
- Wannan Medical College Yijishan Hospital, Wuhu, Anhui, China

REFERENCES:
- [Derived] Hu H, Ma F, Gong L, Wang Y, Xu M, Sun H, Hu Q, Wang P, Han L, Xie H. Immunogenicity and safety of a recombinant Omicron BA.4/5-Delta COVID-19 vaccine ZF2202-A in Chinese adults. Vaccine. 2024 May 31;42(15):3522-3528. doi: 10.1016/j.vaccine.2024.04.058. Epub 2024 May 3. PMID 38704251
- [Derived] He Q, An Y, Zhou X, Xie H, Tao L, Li D, Zheng A, Li L, Xu Z, Yu S, Wang R, Hu H, Liu K, Wang Q, Dai L, Xu K, Gao GF. Neutralization of EG.5, EG.5.1, BA.2.86, and JN.1 by antisera from dimeric receptor-binding domain subunit vaccines and 41 human monoclonal antibodies. Med. 2024 May 10;5(5):401-413.e4. doi: 10.1016/j.medj.2024.03.006. Epub 2024 Apr 3. PMID 38574739